CLINICAL TRIAL: NCT01152554
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled, Phase III, Long-Term Safety and Tolerability Study of TC-5214 (S-mecamylamine) as an Adjunct to an Antidepressant in Patients With Major Depressive Disorder Who Exhibit an Inadequate Response to Antidepressant Therapy
Brief Title: A Study to Assess the Long- Term Safety of TC-5214 as an Adjunct Therapy in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4130C00007
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Results first posted 2012-10-29 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Major Depressive Disorder; MDD; Depression
Keywords: Major Depressive Disorder; MDD; Depression; Safety; add-on therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SSRI/Serotonin/SNRI + TC-5214 1-4 mg (Experimental): Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + TC-5214 1-4 mg BID
  Interventions: Drug: TC-5214
- SSRI/Serotonin/SNRI + placebo (Placebo Comparator): Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-5214 — Tablet, oral, twice daily for 52 weeks
  Arms: SSRI/Serotonin/SNRI + TC-5214 1-4 mg
Drug: Placebo — Tablet, oral, twice daily for 52 weeks
  Arms: SSRI/Serotonin/SNRI + placebo

SUMMARY:
The purpose of this study is to determine if TC-5214 or placebo (a tablet that looks like medicine tablet or capsule, but contains no active medicine) is safe and effective when taken for 52 weeks with another antidepressant medicine.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent before initiation of any study-related procedures.
* The patient must have a clinical diagnosis of major depressive disorder (MDD) with inadequate response to no more than one antidepressant.
* Outpatient status at enrollment and randomization.

Exclusion Criteria:

* Patients with a lifetime history of bipolar disorder, psychotic disorder or post-traumatic stress disorder.
* Patients with a history of suicide attempts in the past year and/or seen by the investigator as having a significant history of risk of suicide or homicide.
* Patients with significant liver, kidney, lung, heart, neurological, or any other medical conditions that might confound the study or put the patient at greater risk during study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 813 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans A. Eriksson, MD, Ph.D, MBA, Study Director — AstraZeneca; Andrew . J Cutler, MD, Principal Investigator — Florida Clinical Research Center, LLC
Locations (94):
- United States (93):
  - Research Site, Birmingham, Alabama
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Arcadia, California
  - Research Site, Beverly Hills, California
  - Research Site, Carson, California
  - Research Site, Cerritos, California
  - Research Site, Chino, California
  - Research Site, Costa Mesa, California
  - Research Site, Encino, California
  - Research Site, Escondido, California
  - Research Site, Garden Grove, California
  - Research Site, Irvine, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Pico Rivera, California
  - Research Site, Riverside, California
  - Research Site, Sherman Oaks, California
  - Research Site, Torrance, California
  - Research Site, Upland, California
  - Research Site, Denver, Colorado
  - Research Site, Norwalk, Connecticut
  - Research Site, Norwich, Connecticut
  - Research Site, Bradenton, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Maitland, Florida
  - Research Site, North Miami, Florida
  - Research Site, Orange City, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pinecrest, Florida
  - Research Site, Plantation, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Roswell, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Schaumburg, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Lafayette, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Prairie Village, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Florence, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Gaithersburg, Maryland
  - Research Site, Glen Burnie, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Weymouth, Massachusetts
  - Research Site, Flowood, Mississippi
  - Research Site, Creve Coeur, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Toms River, New Jersey
  - Research Site, Willingboro, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Fresh Meadows, New York
  - Research Site, Mount Kisco, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Staten Island, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Beechwood, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Mason, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Jenkintown, Pennsylvania
  - Research Site, Norristown, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Friendswood, Texas
  - Research Site, Irving, Texas
  - Research Site, Lake Jackson, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Woodstock, Vermont
  - Research Site, Seattle, Washington
  - Research Site, South Kirkland, Washington
  - Research Site, Middleton, Wisconsin
- Research Site, San Juan, Puerto Rico

REFERENCES:
- [Derived] Tummala R, Desai D, Szamosi J, Wilson E, Hosford D, Dunbar G, Eriksson H. Safety and tolerability of dexmecamylamine (TC-5214) adjunct to ongoing antidepressant therapy in patients with major depressive disorder and an inadequate response to antidepressant therapy: results of a long-term study. J Clin Psychopharmacol. 2015 Feb;35(1):77-81. doi: 10.1097/JCP.0000000000000269. PMID 25514064
- See also: CSR-D4130C00007.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=337&filename=CSR-D4130C00007.pdf
- See also: D4130C00007/Clinical Study Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=337&filename=D4130C00007_Revised_CSP_1_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in the US between 22 June 2010 and 07 February 2012.
Pre-assignment Details: The study had an up to 21-day screening/washout period, and an 6-week prospective open-label antidepressant treatment (ADT) period to identify the target patient population of inadequate responders to ADT (a HAMD-17 total score of ≥10 and a CGI-S score ≥3).
Groups:
- TC-5214: Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + TC-5214, 1-4 mg BID
- Placebo: Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + Placebo BID
Period: Overall Study
Arm/Group | TC-5214 | Placebo
Started | 610 | 203
Received Treatment | 607 | 201
Completed | 276 | 92
Not Completed | 334 | 111
Not completed — Withdrawal by Subject | 73 | 28
Not completed — Eligiblity criteria not fulfilled | 0 | 1
Not completed — Adverse Event | 67 | 14
Not completed — Severe non-compliance to protocol | 36 | 14
Not completed — Condition under investigation worsened | 5 | 2
Not completed — Lack of Efficacy | 20 | 3
Not completed — Study-specific withdrawal criteria | 17 | 8
Not completed — Lost to Follow-up | 87 | 32
Not completed — Other | 28 | 8
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TC-5214 | Placebo | Total
Number analyzed (Participants) | 610 | 203 | 813
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (11.68) | 42.8 (11.75) | 43.1 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 418 | 148 | 566
  Male | 192 | 55 | 247
Race/Ethnicity, Customized [Number; unit: participants]
  White | 467 | 149 | 616
  Black or African American | 121 | 44 | 165
  Asian | 10 | 4 | 14
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  American Indian or Alaska Native | 0 | 2 | 2
  Other | 11 | 4 | 15
Hamilton Rating Scale for Depression-17 items (HAMD-17) total score at randomization [Mean (Standard Deviation); unit: Scores on a scale] — A 17-item, clinician-rated scale that assesses depressive symptoms. The HAMD-17 consists of 17 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The HAMD-17 total score is calculated as the sum of the 17 individual symptom scores; the total score can range from 0 to 52. Higher HAMD-17 scores indicate more severe depression.
  Scores on a scale | 18.4 (4.49) | 18.6 (4.61) | 18.5 (4.52)
Montgomery-Asberg Depression Rating Scale (MADRS) total score at randomization [Mean (Standard Deviation); unit: Scores on a scale] — A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
  Scores on a scale | 23.5 (6.34) | 23.4 (5.85) | 23.4 (6.21)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Patients Experiencing at Least One Adverse Event (AE)
Description: The frequency of patients experiencing at least one AE during the randomized treatment or follow-up periods was calculated.
Time Frame: Randomization (Week 0) to end of the follow-up period (Week 54)
Population: Safety analysis set including all randomized patients who received at least 1 dose of investigational product (TC-5214 or placebo) and for whom any postdose data were available.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | TC-5214 | Placebo
Number analyzed (Participants) | 607 | 201
percentage of participants analyzed | 82.4 | 84.6

2. Primary Outcome: Frequency of Patients Experiencing AEs That Resulted in Discontinuation of Investigational Product (IP)
Description: The frequency of patients experiencing AEs that resulted in discontinuation of IP during the randomized treatment or follow-up periods was calculated.
Time Frame: Randomization (Week 0) to end of the follow-up period (Week 54)
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Arm/Group | TC-5214 | Placebo
Number analyzed (Participants) | 607 | 201
percentage of participants analyzed | 10.5 | 7.0

3. Primary Outcome: Frequency of Patients Experiencing Serious Adverse Events (SAEs)
Description: The frequency of patients experiencing serious adverse events (SAEs) during the randomized treatment or follow-up periods was calculated.
Time Frame: Randomization (Week 0) to end of the follow-up period (Week 54)
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Arm/Group | TC-5214 | Placebo
Number analyzed (Participants) | 607 | 201
percentage of participants analyzed | 3.6 | 2.5

4. Secondary Outcome: Sustained Efficacy at 3 Months, Defined as a Montgomery-Asberg Depression Rating Scale (MADRS) Total Score of ≤12 at Week 12 and All Visits up to and Including Week 24
Description: The percentage of patients with a a MADRS total score of ≤12 at Week 12 and all visits up to and including Week 24 was calculated. One intermediate occurrence of a MADRS total score >12 but ≤16 or missing was allowed from Week 16 to Week 20.
  A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Week 12 to Week 24
Population: Modified intent-to-treat analysis set including all randomized patients who received at least 1 dose of investigational product (TC-5214 or placebo) and who had a total MADRS score at randomization and a total HAMD-17 score ≥16 and a CGI-S score ≥4 at randomization.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | TC-5214 | Placebo
Number analyzed (Participants) | 391 | 136
percentage of participants analyzed | 18.2 | 20.6
Statistical Analysis 1: Comparison: TC-5214 vs Placebo; Logistic regression model including treatment and pooled center as fixed effects and the randomization MADRS total score as a covariate; Test type: Superiority or Other; p = 0.697, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.54 to 1.50], Standard Error of Mean 0.24 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

5. Secondary Outcome: Sustained Efficacy at 9 Months, Defined as a MADRS Total Score of ≤12 at Week 12 and at All Visits up to and Including Week 52
Description: The percentage of patients with a MADRS total score of ≤12 at Week 12 and at all visits up to and including Week 52 was calculated. Two intermediate occurrences (not consecutive) of a MADRS >12 but ≤16 or missing were allowed from Week 16 to Week 48.
  A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Week 12 to Week 52
Population: as for outcome 4
Measure: Number; unit: percentage of patients analyzed
Arm/Group | TC-5214 | Placebo
Number analyzed (Participants) | 391 | 136
percentage of patients analyzed | 9.7 | 12.5
Statistical Analysis 1: Comparison: TC-5214 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.582, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.45 to 1.57], Standard Error of Mean 0.27 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

6. Secondary Outcome: Change in the Clinician-rated Global Outcome of Severity as Measured by the Clinical Global Impression-Severity (CGI-S) Score From Randomization (Week 0) to End of Treatment (Week 52)
Description: A 3-part, clinician-administered scale that rates the improvement or worsening of the patient's illness from randomization (baseline). Each item is scored on a 1 to 7 scale. Higher CGI-S scores indicate greater illness severity.
Time Frame: Randomization (Week 0) to end of treatment (Week 52)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TC-5214 | Placebo
Number analyzed (Participants) | 176 | 68
units on a scale | -1.8 (1.17) | -1.6 (1.17)

7. Secondary Outcome: Change in Functional Impairment From Randomization (Week 0) to End of Treatment (Week 52) as Measured by the Sheehan Disability Scale (SDS) Total Score
Description: Sheehan Disability Scale (SDS) is 5-item, self-administered scale that measures the extent a patient is impaired by their disease. Higher scores indicate more severe impairment. The SDS total score is calculated as the sum of the score for the 3 inter-correlated domains (school/work, social life, and family life/home responsibilities) and ranges from 0 (unimpaired) to 30 (highly impaired).
Time Frame: Randomization (Week 0) to end of treatment (Week 52)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TC-5214 | Placebo
Number analyzed (Participants) | 185 | 70
units on a scale | -6.98 (7.909) | -7.44 (7.530)

8. Secondary Outcome: Change in Overall Quality of Life and Satisfaction From Randomization (Week 0) to End of Treatment (Week 52) by Assessing the Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) % Maximum Total Score
Description: The Q-LES-Q-SF total score is derived by summing item scores 1 to 14. Higher scores are indicative of greater enjoyment or satisfaction in each domain. The Q-LES-Q-SF % maximum total score is calculated as 100% × (Q-LES-Q-SF total score - 14) / 56, and can range from 0% to 100%.
Time Frame: Randomization (Week 0) to end of treatment (Week 52)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TC-5214 | Placebo
Number analyzed (Participants) | 184 | 70
units on a scale | 10.83 (18.744) | 11.62 (17.006)

9. Secondary Outcome: Change in EuroQol - 5 Dimensions (EQ-5D) From Randomization (Week 0) to End of Treatment (Week 52)
Description: A self-assessment questionnaire that provides 2 measures of health status. The EQ-5D index score is a weighted linear combination over 5 dimensions of health status. The score for each of the 5 dimensions can range from 1 to 3, and an equation is used to calculate the EQ-5D index score. The EQ-5D index score can range from possible negative values to a maximum of 1.0. The EQ-VAS is a visual analog scale with a range of 0 to 100. For both variables, a higher score indicates a better health state.
Time Frame: Randomization (Week 0) to end of treatment (Week 52)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TC-5214 | Placebo
Number analyzed (Participants) | 177 | 68
units on a scale
  EQ-5D index score | 0.081 (0.2021) | 0.071 (0.1500)
  EQ-5D VAS score | 8.7 (20.04) | 11.9 (21.06)

ADVERSE EVENTS:
Groups:
- Placebo: Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + Placebo
Arm/Group | Placebo | TC-5214
Serious Adverse Events (participants affected / at risk) | 5/201 | 22/607
Other Adverse Events (participants affected / at risk) | 151/201 | 451/607
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=201) | TC-5214 (N=607)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Oral Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Brain Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 2 (2)
Ovarian Torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=201) | TC-5214 (N=607)
Constipation (Gastrointestinal disorders) | 12 (14) | 120 (147)
Diarrhoea (Gastrointestinal disorders) | 20 (23) | 65 (80)
Nausea (Gastrointestinal disorders) | 24 (27) | 64 (79)
Dry Mouth (Gastrointestinal disorders) | 10 (11) | 59 (61)
Vomiting (Gastrointestinal disorders) | 13 (21) | 32 (40)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 12 (12)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 14 (16)
Flatulence (Gastrointestinal disorders) | 4 (4) | 14 (15)
Abdominal Distension (Gastrointestinal disorders) | 4 (5) | 5 (5)
Fatigue (General disorders) | 17 (18) | 39 (43)
Seasonal Allergy (Immune system disorders) | 5 (5) | 11 (12)
Upper Respiratory Tract Infection (Infections and infestations) | 30 (39) | 104 (122)
Nasopharyngitis (Infections and infestations) | 22 (26) | 59 (70)
Sinusitis (Infections and infestations) | 11 (14) | 28 (32)
Urinary Tract Infection (Infections and infestations) | 10 (11) | 26 (30)
Influenza (Infections and infestations) | 7 (8) | 19 (22)
Bronchitis (Infections and infestations) | 5 (5) | 12 (12)
Gastroenteritis (Infections and infestations) | 5 (6) | 14 (14)
Gastroenteritis Viral (Infections and infestations) | 5 (5) | 13 (13)
Contusion (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Muscle Strain (Injury, poisoning and procedural complications) | 4 (4) | 7 (7)
Weight Increased (Injury, poisoning and procedural complications) | 14 (14) | 27 (27)
Blood Pressure Increased (Injury, poisoning and procedural complications) | 5 (6) | 8 (9)
Increased Appetite (Metabolism and nutrition disorders) | 5 (5) | 11 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 26 (35)
Back Pain (Musculoskeletal and connective tissue disorders) | 18 (21) | 20 (23)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 15 (16)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 13 (13)
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 11 (11)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 9 (11)
Headache (Nervous system disorders) | 34 (52) | 102 (170)
Dizziness (Nervous system disorders) | 16 (24) | 75 (99)
Dizziness Postural (Nervous system disorders) | 3 (3) | 28 (43)
Somnolence (Nervous system disorders) | 9 (9) | 31 (33)
Sedation (Nervous system disorders) | 4 (4) | 12 (12)
Memory Impairment (Nervous system disorders) | 4 (4) | 5 (6)
Migraine (Nervous system disorders) | 5 (5) | 8 (8)
Paraesthesia (Nervous system disorders) | 5 (6) | 7 (7)
Tremor (Nervous system disorders) | 4 (4) | 5 (5)
Insomnia (Psychiatric disorders) | 18 (20) | 47 (52)
Abnormal Dreams (Psychiatric disorders) | 7 (7) | 28 (29)
Agitation (Psychiatric disorders) | 5 (6) | 21 (22)
Anxiety (Psychiatric disorders) | 1 (1) | 15 (17)
Bruxism (Psychiatric disorders) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 15 (15)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 11 (12)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 13 (13)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5) | 17 (19)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
Hypertension (Vascular disorders) | 9 (9) | 15 (15)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days